CLINICAL TRIAL: NCT00031278
Title: A Phase I/II Open Label, Multi-Center Study For The Evaluation Of The Combination Of CpG 7909 And Herceptin® In Patients With Metastatic Breast Cancer
Brief Title: Safety And Efficacy Study Of The Combination Of CpG 7909 And Herceptin In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C005; C005; A8501020
Record Dates: First submitted 2002-02-28; First posted 2002-03-01 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Carcinoma, Metastatic Breast
Keywords: Metastatic; Breast; Cancer; immunotherapy; CPG 7909
MeSH Terms: conditions — Carcinoma; Neoplasm Metastasis; Neoplasms | interventions — ProMune; Trastuzumab

ARMS (4):
- Cohort 1 (Experimental): 0.01 mg/kg CPG 7909 plus Herceptin®
  Interventions: Drug: CPG 7909; Drug: Herceptin®
- Cohort 2 (Experimental): 0.04 mg/kg CPG 7909 plus Herceptin®
  Interventions: Drug: CPG 7909; Drug: Herceptin®
- Cohort 3 (Experimental): 0.16 mg/kg CPG 7909 plus Herceptin®
  Interventions: Drug: CPG 7909; Drug: Herceptin®
- Cohort 4 (Experimental): 0.32 mg/kg CPG 7909 plus Herceptin®
  Interventions: Drug: CPG 7909; Drug: Herceptin®

INTERVENTIONS:
Drug: CPG 7909 — Each 0.01 mg/kg CPG 7909 treatment will consist of a monitored 2-hour infusion given once weekly until disease progression or a maximum of 24 weeks.
  Other Names: PF-3512676, ProMune
  Arms: Cohort 1
Drug: Herceptin® — Herceptin® will be administered at a dose of 2 mg/kg IV according to the Herceptin® package insert
  Other Names: trastuzumab
  Arms: Cohort 1
Drug: CPG 7909 — Each 0.04 mg/kg CPG 7909 treatment will consist of a monitored 2-hour infusion given once weekly until disease progression or a maximum of 24 weeks.
  Other Names: PF-3512676, ProMune
  Arms: Cohort 2
Drug: Herceptin® — Herceptin® will be administered at a dose of 2 mg/kg IV according to the Herceptin® package insert
  Other Names: trastuzumab
  Arms: Cohort 2
Drug: CPG 7909 — Each 0.16 mg/kg CPG 7909 treatment will consist of a monitored 2-hour infusion given once weekly until disease progression or a maximum of 24 weeks.
  Other Names: PF-3512676, ProMune
  Arms: Cohort 3
Drug: Herceptin® — Herceptin® will be administered at a dose of 2 mg/kg IV according to the Herceptin® package insert
  Other Names: trastuzumab
  Arms: Cohort 3
Drug: CPG 7909 — Each 0.32 mg/kg CPG 7909 treatment will consist of a monitored 2-hour infusion given once weekly until disease progression or a maximum of 24 weeks.
  Other Names: PF-3512676, ProMune
  Arms: Cohort 4
Drug: Herceptin® — Herceptin® will be administered at a dose of 2 mg/kg IV according to the Herceptin® package insert
  Other Names: trastuzumab
  Arms: Cohort 4

SUMMARY:
The purpose of this study is to determine if the combination of CPG 7909 and Herceptin is safe and effective in the treatment of metastatic breast cancer.

RATIONALE: There is preclinical data that supports the hypothesis that CPG 7909 may potentiate the action of Herceptin. This Phase I/II study is designed to evaluate the safety and efficacy of the combination treatment of CPG 7909 and Herceptin in patients with metastatic breast cancer who have previously been treated with Herceptin and chemotherapy.

SCHEDULE: Patients will receive CPG 7909 weekly for up to six months.

DETAILED DESCRIPTION:
Phase II part of study not initiated because the development plan modified the route of administration to subcutaneous injection.

ELIGIBILITY:
INCLUSION CRITERIA Inclusion Criteria

* Histologically confirmed breast cancer with metastases.
* Tumor that has overexpression of HER2 as documented by being either FISH-positive or HER2/neu 3+ confirmed by immunohistochemistry.
* Patients must be candidates for single agent Herceptin treatment according to the Herceptin® label.

Exclusion Criteria

* Any prior therapy with anthracycline + Herceptin®.
* Significant cardiovascular disease (e.g., NYHA class 3 congestive heart failure, myocardial infarction within the past 6 months, unstable angina; coronary angioplasty within the past 6 months, uncontrolled atrial or ventricular cardiac arrhythmias) or left ventricular ejection fraction < 50%.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Phase I: To evaluate the safety, tolerability and and MTD of several dose levels of CPG 7909 of CPG 7909 in combination with the standard Herceptin® treatment in patients with metastatic breast cancer
Phase II: Evaluate tumor response and safety of CPG 7909 in combination with Herceptin® in patients with metastatic breast cancer

SECONDARY OUTCOMES:
Phase I: To evaluate tumor response, duration of response, time to disease progression, and survival time
Phase II: To evaluate duration of response, time to disease progression, and survival time

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, M.D., Ph.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Univ. of Connecticut Health Center, Farmington, Connecticut
  - Cancer Research Network, Inc., Plantation, Florida
  - Greenebaum Cancer Center at Univ. of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Center, University of Michigan, Ann Arbor, Michigan
  - Cancer Center at Saint Barnabas Medical Center, Livingston, New Jersey
  - Univ. of Pittsburgh Cancer Institute, Magee Women's Hosp., Pittsburgh, Pennsylvania
  - Fletcher Allen Health Care, Burlington, Vermont